CLINICAL TRIAL: NCT05018390
Title: Impact of Osteopathic Manipulative Treatment on External Lateral Ocular Pursuit, Measured in Healthy Human Adults: a Randomized, Double-blind, Controlled Study
Brief Title: Impact of Osteopathic Manipulative Treatment on Pursuit Eye Movements in Healthy Human Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ecole d'ostéopathie de Paris (Other)
Collaborators: University of Paris 5 - Rene Descartes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OSTEOM-1
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Healthy
Keywords: Osteopathic manipulative treatment; Ocular pursuit
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The practitioner providing the actual OMT or sham Treatment will not be involved in collecting eye movement data. The persons collecting eye movement data will not know the group to which participants will have been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OMT (Experimental): Osteopathic manipulative treatment : participants will receive low-amplitude tissue mobilizations on peripheral, vertebral, cranial and/or visceral articular systems.
  Interventions: Other: Osteopathic manipulative treatment
- Sham (Sham Comparator): Participants will be applied gestures that look like actual osteopathic manipulations but are not therapeutic.
  Interventions: Other: Sham Osteopathic manipulative treatment
- Test-retest (No Intervention): Participants will undergo the two eye movement measurements, but will not receive any (actual or sham) treatment. 30 minutes will elapse between the two measurements.

INTERVENTIONS:
Other: Osteopathic manipulative treatment — Participants will be positioned on an exam table supine, seated, or decubitus. Osteopathic manipulations will consist in corrective micro-movements applied on synovial joints, on the skull, the teeth and/or visceral structures of the abdomen or the thorax. Local pressures won't exceed a few tens of grams/cm². Practitioners will realize between 15 and 25 technical gestures per participant. Treatment will last 30 minutes (plus or minus 5 minutes) on average. The technical gestures are referenced in the Glossary of Osteopathic Terminology published by the American Association of Colleges of Osteopathic Medicine (2017).
  Arms: OMT
Other: Sham Osteopathic manipulative treatment — Participants will be positioned on an exam table supine, seated, or decubitus. They will receive 20 gestures that will be standardized and different from actual osteopathic manipulations (but not identifiable as sham manipulations by the participants). The duration of the sham treatment will be the same as the actual treatment.
  Arms: Sham

SUMMARY:
The idea that osteopathic manipulative treatments (OMTs) should have an impact on the human visual system is not new. Nevertheless, there is a lack of scientific, objective, and experimental evidence. Our goal is to conduct a randomized, double-blind, controlled study to evaluate the effect of OMT on ocular pursuit. Eye movements will be measured by an infra-red video-based eye tracking system with a high spatial and temporal resolution. OMTs will be similar to regular treatments given by osteopaths in their daily practice. We hypothesize that OMT will improve the quality of ocular pursuit.

DETAILED DESCRIPTION:
Our hypothesis is based on the implication of the fascial system (i.e., connective tissues) in the structural continuity that gives form and function to every tissue and organ. Fascial tissue, on which osteopathic manipulations are acting by restoring its elasticity, is also present in the eye cavity. The connection between fascia might explain how osteopathic manipulations, applied on structures which can be far from the original dysfunctional point, might improve oculomotricity.

Before and after OMT, practitioners will estimate the lateral and medial oculomotor muscles' and the fascia's tissue elasticity with a manual test. They will softly mobilize the eyeballs in medial and lateral directions (the amplitude of these passive mobilizations will always be lower than active eye rotations) and give an elasticity score. Before and after these tests, pursuit eye movements will be recorded by an independent technician. Participants will be asked to track a target that will be displaced horizontally on a computer screen. The target will move 30 times from left to right and 30 times from right to left with a constant speed of 20 degrees of visual angle per second.

The study will involve three independent groups (experimental, sham, test-retest) of healthy participants. We expect that pursuit improvement will be larger in the experimental group than in the two other groups. Moreover, as secondary goals, we will evaluate the correlation between pursuit eye movement data (obtained with a technical device, in a standardized situation) and subjective assessments of oculomotor muscles' elasticity made by the practitioners providing OMTs. We will also examine the possible practitioner effect (two exclusive osteopaths will provide OMTs).

ELIGIBILITY:
Inclusion Criteria:

* Adult between 18 and 35 years of age
* Affiliated to the French Social Security scheme
* Ability to understand and sign the written consent form

Exclusion Criteria:

* Eye movements that cannot be calibrated correctly and therefore measured by the eye-tracker
* Visual deficit that prevents from performing the ocular task
* Pregnancy or breastfeeding
* Neurologic, psychiatric or epileptic disorder, or any other neuromuscular disorder
* Medical treatment affecting the central, autonomous or peripheral nervous system, or affecting vigilance and/or attention
* Skull fracture less than 12 months ago, symptomatic whiplash less than 3 months ago, spinal pain, fever, abdominal or pelvic pain, myopathy, ocular pain, or nystagmus
* Legal protection
* Major risk to develop severe corona virus disease illness, or living with people presenting such a risk

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Duration of external lateral ocular pursuit | immediately before treatment
  Time spent to track a moving target, by generating smooth eye movements (as opposed to ocular saccades) with a velocity close to the target velocity. Metric: millisecond.
Mean change from baseline in duration of external lateral ocular pursuit | immediately after treatment
  Change from baseline in time spent to track a moving target, by generating smooth eye movements (as opposed to ocular saccades) with a velocity close to the target velocity. Metric: millisecond.
Reaction time | immediately before treatment
  Time elapsed between target displacement initiation and ocular pursuit initiation. Metric: millisecond.
Mean change from baseline in reaction time | immediately after treatment
  Mean change from baseline in time elapsed between target displacement initiation and ocular pursuit initiation. Metric: millisecond.

SECONDARY OUTCOMES:
Score on the test of eyeball passive manual mobilization | immediately before treatment
  Tissue elasticity of an oculomotor muscle will be assessed using a 3-points scale (1 = no resistance to the mobilization, 3 = strong resistance). Four muscles (two per eyeball) will be assessed. Maximal score = 12 points.
Score on the test of eyeball passive manual mobilization | immediately after treatment
  Tissue elasticity of an oculomotor muscle will be assessed using a 3-points scale (1 = no resistance to the mobilization, 3 = strong resistance). Four muscles (two per eyeball) will be assessed. Maximal score = 12 points.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Gharmaoui, MD, Principal Investigator — Ecole d'Osteopathie de Paris
Locations (1):
- Ecole d'Osteopathie de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bordoni B, Zanier E. Clinical and symptomatological reflections: the fascial system. J Multidiscip Healthc. 2014 Sep 18;7:401-11. doi: 10.2147/JMDH.S68308. eCollection 2014. PMID 25258540